CLINICAL TRIAL: NCT00142285
Title: Efficacy of Zinc in the Treatment of Outpatient Pneumonia in an Urban Slum Among Children Less Than 2 Years Old
Brief Title: Zinc Pneumonia Outpatient Trial in Children < 2 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-010
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2006-07

CONDITIONS: Pneumonia
Keywords: pneumonia; zinc; treatment; efficacy; children
MeSH Terms: conditions — Pneumonia | interventions — Zinc Sulfate

INTERVENTIONS:
Drug: Zinc sulphate (20 mg)

SUMMARY:
The purpose of this study is to determine whether zinc can be used in combination with standard antibiotics to reduce the duration of illness and the likelihood of treatment failure among children less than two years old who have non-severe, outpatient pneumonia.

DETAILED DESCRIPTION:
This study is a follow up to an earlier study among hospitalised children less than two years old with severe pneumonia who were administered zinc as an adjuvant along with standard antimicrobial agents. That study found a 20% reduction in illness duration and hospitalisation, as well as a 3 - 9 fold reduction in treatment failure for children given zinc along with standard antimicrobial management. However, since most pneumonia is managed in an outpatient setting, it is important to know if it works in this setting as well. We hypothesise that zinc may act as an acute phase reactant in the early stages of outpatient non-severe pneumonia to reduce both the duration of illness and the likelihood of treatment failure.

To test this, we will randomise children less than two years old to receive either zinc or placebo can as an adjuvant to standard oral antimicrobial agents in the acute treatment of non-severe pneumonia in an outpatient urban setting. Oral antibiotics will be given for a standard five-day course, while zinc (20 mg) or placebo will be administered once-daily for 10 days. Patients will be followed up on a daily basis at home to monitor their progress and document compliance.

Outcomes will be a comparison between zinc and placebo groups on duration of illness, as measured by specific signs of pneumonia, and treatment failure, as measured by change of antibiotics or hospitalisation for failure to improve or worsening condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pneumonia

Exclusion Criteria:

* Wheezing at presentation History of chronic lung, heart or other system disease suspected tuberculosis, active measles, severe malnutrition requiring hospitalisation, signs of systemic illness (sepsis, meningitis), those who have already received zinc/placebo supplements during this study, those known to be pre-treated with antibiotics prior to presenting to clinic

Ages: 1 Week to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2260 (Estimated)
Dates: Start 2004-11; Primary Completion 2006-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Duration of illness
Treatment failure

SECONDARY OUTCOMES:
Incidence of subsequent illness episodes (pneumonia and any other)

CONTACTS AND LOCATIONS:
Overall Officials: W. Abdullah Brooks, MD, MPH, Principal Investigator — ICDDR,B: Centre for Health & Population Research
Locations (1):
- Kamalapur Urban Site, ICDDR,B: Centre for Health & Population Research, Dhaka, Bangladesh

REFERENCES:
- [Background] Brooks WA, Yunus M, Santosham M, Wahed MA, Nahar K, Yeasmin S, Black RE. Zinc for severe pneumonia in very young children: double-blind placebo-controlled trial. Lancet. 2004 May 22;363(9422):1683-8. doi: 10.1016/S0140-6736(04)16252-1. PMID 15158629
- See also: Link to ICDDR,B, then click on 'Publications' or 'Programmes and themes' — http://www.icddrb.org